CLINICAL TRIAL: NCT03223844
Title: Disentangling Pre- and Postsynaptic Aspects of Amphetamine-induced Sensitization: a Combined [18F]DOPA / [11C]-(+)-PHNO PET Study
Brief Title: Influence of Amphetamine-induced Sensitization on Dopamine Synthesis and Release
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ana Weidenauer, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16969
Record Dates: First submitted 2017-07-08; First posted 2017-07-21 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Schizophrenia; Psychosis; Sensitisation
Keywords: Dopamine; Amphetamine; Positron Emission Tomography; Magnetic Resonance Imaging; Schizophrenia; Psychosis; [18F]FDOPA; [11C]-(+)-PHNO
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Dextroamphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Experimental): Measurement of Dextroamphetamine Sulfate-induced dopamine release and synthesis before and after amphetamine sensitization.
  Interventions: Drug: Dextroamphetamine Sulfate

INTERVENTIONS:
Drug: Dextroamphetamine Sulfate — Repeated oral administration of dexamphetamine 0.4mg/KG bodyweight four times.
  Other Names: [11C]-(+)-PHNO PET, [18F]FDOPA PET

SUMMARY:
Patients with schizophrenia show enhanced dopamine synthesis capacity and release, an effect that can be evoked in healthy subjects by repeated amphetamine administration. Therefore for the first time the relationship between dopamine synthesis and release will be studied in healthy subjects before and after amphetamine sensitization in order to better understand adaptive mechanisms of the dopamine system.

DETAILED DESCRIPTION:
Positron emission tomography (PET) studies have consistently shown increased brain dopamine (DA) synthesis and enhanced d-amphetamine-induced DA release in patients with schizophrenia. Repeated administration of d-amphetamine leads to an increased subjective and behavioral drug-response. This effect, termed "sensitization", is paralleled by an increase in dopamine release to levels akin to those observed in schizophrenia. Schizophrenia thus goes along with a state of 'natural sensitization' towards amphetamines. However, while it is known that DA synthesis and release are both enhanced in schizophrenia, it is unknown whether sensitization changes indices of presynaptic DA synthesis in the striatum of healthy subjects. Thus, for the first time, this project will study the effects of repeated d-amphetamine on uptake of the DA precursor [18F]FDOPA and on d-amphetamine-induced changes in binding of the D2/3 receptor agonist radioligand [11C]-(+)PHNO in a within-subject design. Before and after amphetamine sensitization by repeated intermittent administration subjects will receive an [18F]FDOPA and and a [11C]-(+)PHNO PET scan. For the investigation of the influence of functional and structural cortical properties on dopamine synthesis and release, functional and structural magnet resonance imaging will be performed before and after sensitization.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-65, in good general health based on history and physical examination
* Psychiatrically healthy as determined by the Mini-International Neuropsychiatric Interview (M.I.N.I.PLUS) (94))
* No relevant abnormalities in laboratory screening including thyroid function tests, blood cell count, serum electrolytes, liver and kidney function, and urinalysis
* No clinically relevant findings in electrocardiography (ECG)
* No clinically relevant findings in vital signs (blood pressure and pulse)
* No regular use of illegal drugs or alcohol abuse based on declared history and confirmed by urine drug screening
* No history of repeated AMPH (AMPH), cocaine or other stimulant drug use

Exclusion Criteria:

* Evidence of present psychiatric or neurological illness according to M.I.N.I.-Plus (any personal or first-degree relative history of: schizophrenia, bipolar disorder, attention-deficit/hyperactivity disorder, and substance dependence)
* Recreational use of psychostimulant drugs in the past two years; lifetime use of psychostimulants exceeding five exposures
* Medically significant biochemical or hematological abnormality on screening laboratory studies
* Women of childbearing potential: Current pregnancy or breast-feeding
* Clinically relevant abnormalities in the electro-cardiogram (ECG)
* History of myocardial infarction or angina pectoris
* Positive urine drug screen within one week prior to PET study day
* Presence of ferromagnetic metal in the body or heart pacemaker
* Claustrophobia
* Any history of arterial hypertension or paroxysmal hypertensive states
* Established diagnosis of advanced arteriosclerosis
* Established diagnosis of hyperthyroidism
* History of hypersensitivity to sympathomimetics
* History of head trauma resulting in loss of consciousness that required medical intervention
* Lifetime history of substance dependence (except nicotine)
* If participation in this study would exceed the annual radiation dose limits (30 mSv) for human subjects
* Subjects currently participating in research studies
* Suicidal ideation or likelihood of a suicide or homicide attempt

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
[18F]FDOPA Ki values | Baseline and 2 weeks after amphetamine sensitization, Week 1 and Week 4
  Relative change in regional [18F]FDOPA Ki values after AMPH sensitization

SECONDARY OUTCOMES:
[11C]-(+)-PHNO BPND values | Baseline and 2 weeks after amphetamine sensitization, Week 1 and Week 4
  Relative change in regional [11C]-(+)-PHNO BPND values after AMPH administration before and after sensitization
Subjective ratings of amphetamine effects (Drug Effects Questionnaire) | Baseline, after i.v. amphetamine during PHNO PET, on each of the two sensitization visits and 2 weeks after amphetamine sensitization during PHNO PET scanning over the course of 4 weeks. Time points: Week 1 Week 2 Week 4
  Subjective ratings will be assessed via questionnaire (Drug Effects Questionnaire) four times throughout the study.
Subjective ratings of amphetamine effects (Subjective States Questionnaire) | Baseline, after i.v. amphetamine during PHNO PET, on each of the two sensitization visits and 2 weeks after amphetamine sensitization during PHNO PET scanning over the course of 4 weeks. Time points: Week 1 Week 2 Week 4
  Subjective ratings will be assessed via questionnaire (Subjective States Questionnaire) four times throughout the study.
Cognitive measures | At baseline, on each of the two sensitization visits after amphetamine administration and 2 weeks after amphetamine sensitization before FDOPA scanning, total timeframe 4 weeks, Time points: Week 1 Week 2 Week 4
  Working memory, reward processing and impulsivity will be assessed via a computerized test battery four times throughout the study
Impulsiveness | Baseline, Week 1
  The personality traits impulsiveness will be assessed once during study participation by the questionnaire Barrat Impulsiveness Scale (BIS).
Personality-related markers | Baseline, Week 1
  Personality traits like novelty seeking will be assessed once during study participation using the Temperament and Character Inventory (TCI).
Peripheral markers of sensitization | Baseline FDOPA scan, baseline PHNO + amphetamine scan, post-sensitization PHNO+ amphetamine scan, post-sensitization FDOPA scan, Time points: Week 1 Week 2 Week 4
  Plasma concentration of the dopamine metabolite HVA, glucose and insulin metabolism related parameters (glucose, glucagon, insulin, c-peptide, somatostatin), plasma cocaine and AMPH-regulated transcript (CART) levels will be measured at each PET study day.
Salivary cortisol | Salivary cortisol will be assessed each time amphetamine is administered: At baseline and 30, 60, 90, 145 and 210 minutes after i.v. or oral amphetamine administration.
  Salivary cortisol will be assessed using Salivettes ®.
Fractional anisotropy (diffusion-weighted tensor imaging) of white matter | Before and after amphetamine sensitization, Week 1, Week 5
  Fractional anisotropy of white matter will be measured by means of magnet resonance imaging.
Gray matter volume | Before and after amphetamine sensitization, Week 1, Week 5
  Gray matter volume will be measured by means of magnet resonance imaging. T1 and PD sequences will be recorded.
Functional connectivity | Before and after amphetamine sensitization, Week 1, Week 5
  Functional connectivity between brain regions will be measured by means of magnet resonance imaging during a resting state of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Weidenauer, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weidenauer A, Bauer M, Sauerzopf U, Bartova L, Praschak-Rieder N, Sitte HH, Kasper S, Willeit M. Making Sense of: Sensitization in Schizophrenia. Int J Neuropsychopharmacol. 2016 Dec 31;20(1):1-10. doi: 10.1093/ijnp/pyw081. Print 2017 Jan. PMID 27613293
- [Background] Sauerzopf U, Sacco R, Novarino G, Niello M, Weidenauer A, Praschak-Rieder N, Sitte H, Willeit M. Are reprogrammed cells a useful tool for studying dopamine dysfunction in psychotic disorders? A review of the current evidence. Eur J Neurosci. 2017 Jan;45(1):45-57. doi: 10.1111/ejn.13418. Epub 2016 Oct 19. PMID 27690184